CLINICAL TRIAL: NCT03137719
Title: Infections and Other Complications of Cirrhosis: A Prospective Multi-Center Study
Brief Title: Infections in Hospitalized Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 010-294
Record Dates: First submitted 2017-03-27; First posted 2017-05-03 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-02

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hospitalized cirrhotic patients are at high risk of complications and adverse outcomes. This study aims to determine the current practice and outcomes in these following areas:

1. Community-acquired infections
2. Nosocomial infections
3. Development of second infections
4. Factors predicting ICU care, organ failure, death, and disability
5. Patterns and adequacy of albumin use in infected and non-infected patients
6. Per and post-liver transplant outcomes
7. Quality-assurance and adequacy of management of complications of cirrhosis such as hepatic encephalopathy, variceal bleeding, hyponatremia, and hypernatremia
8. Regional variations in outcomes and therapeutic strategies

ELIGIBILITY:
Inclusion Criteria:

* Male and Female over 18 years of age
* Cirrhosis as diagnosed by either liver histology or a combination of clinical biochemical (low platelets, elevated bilirubin, and/or INR, low albumin) radiologic (nodular liver on ultrasound) and endoscopic (esophageal varices) criteria
* Subject must be able to understand and provide informed consent
* Evaluated in the ER or admitted to the hospital for non-elective reasons

Exclusion Criteria:

* admitted for elective purpose

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized cirrhotic patients
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Frequency, Cause and Outcome of Community-acquired infections | From admission to 1 year post-discharge from the hospital
  Collecting details of infections including type, organism, antibiotic used, length of stay, ICU stay and outcomes
Frequency, Cause, and Outcome of Nosocomial infections | From admission to 1 year post-discharge from the hospital
  Collecting details of infections including type, organism, antibiotic used, length of stay, ICU stay and outcomes
Development of second infections | From admission to 1 year post-discharge from the hospital
  Distinctly different from primary infection
Factors predicting ICU care, organ failure, death, and disability | From admission to 1 year post-discharge from the hospital
  Admission to the ICU and events/outcomes of that subject's admission
Patterns and adequacy of albumin use in infected and non-infected patients | From admission to 1 year post-discharge from the hospital
  IV albumin administration
Quality-assurance and adequacy of management of complications of cirrhosis such as hepatic encephalopathy, variceal bleeding, hyponatremia, and hypernatremia | From admission to 1 year post-discharge from the hospital
  Blood test and other obvious clinical evidence of decompensation
Peri and post-liver transplant outcomes based on physiological parameters | From admission to 1 year post-discharge from the hospital
  Collection of liver transplant donor and recipient information such as blood group, CMV status, post-transplant infections, immunosuppression regimen, and prophylaxis given.
Regional variations in outcomes and therapeutic strategies | From admission to 1 year post-discharge from the hospital
  Comparison of data between sites conducting this study across the United States and Canada